CLINICAL TRIAL: NCT02991521
Title: Can we be FASTeR? A Multicenter Study Utilizing Right Sided Roll to Improve Sensitivity of the FAST Examination
Brief Title: A Study to Improve the FAST Ultrasound Exam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1606-30
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hemoperitoneum
MeSH Terms: conditions — Hemoperitoneum | interventions — Focused Assessment with Sonography for Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FAST examination after Right sided roll (FASTeR) (Experimental): Subjects will have a standard FAST exam, and will then be rolled onto their right side and the FAST exam will be repeated.
  Interventions: Procedure: Fast exam

INTERVENTIONS:
Procedure: Fast exam — Positional change before Fast exam

SUMMARY:
This research study aims to improve the standard exam called Focused Assessment with Sonography in Trauma (FAST). The FAST exam is an ultrasound test used to identify an abdominal bleed. The study will see if having patients roll on their right side improves the FAST exam. Making the FAST exam better can help trauma doctors save the lives of patients with bleeding.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients who present as a Trauma Activation with clinical history or physical signs of blunt abdominal trauma.

Exclusion Criteria:

* Pregnant females
* Prisoners
* Patients with prohibitive right sided chest trauma
* Patients in extremis undergoing salvage maneuvers (chest compressions or emergent surgical intervention) which prevents performance of an ultrasound examination
* Patient who leave against medical advice or are otherwise removed from the medical system before their work up has been completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Pigneri, MD, Principal Investigator
Locations (2):
- United States (2):
  - Robert Packer Hospital, Sayre, Pennsylvania
  - The Guthrie Clinic, Sayre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cibulas Shumway M, Granet J, Solomon RJ, Parreco JP, Lee SK, Pigneri DA; FASTeR Study Group. Using Right-Sided Roll to Improve Reliability of Focused Assessment with Sonography in Trauma: An Eastern Association for the Surgery of Trauma Multicenter Prospective Study. J Am Coll Surg. 2023 Jan 1;236(1):99-104. doi: 10.1097/XCS.0000000000000443. Epub 2022 Dec 15. PMID 36519913
- See also: Using Right-Sided Roll to Improve Reliability of Focused Assessment with Sonography in Trauma: An Eastern Association for the Surgery of Trauma Multicenter Prospective Study — https://journals.lww.com/journalacs/Citation/2023/01000/Using_Right_Sided_Roll_to_Improve_Reliability_of.18.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from June 2016-October 2020 at 8 designated trauma centers across the United States
Pre-assignment Details: All subjects completed traditional FAST examination in the supine position and FASTeR examination regardless of findings on initial FAST examination
Groups:
- FAST Examination After Right Sided Roll (FASTeR): Subjects complete standard FAST then complete FAST examination after Right sided roll (FASTeR)
Period: Overall Study
Arm/Group | FAST Examination After Right Sided Roll (FASTeR)
Started | 182
Completed | 182
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FAST Examination After Right Sided Roll (FASTeR)
Number analyzed (Participants) | 182
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [38 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 122
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Screening Positive for Blood Around the Abdominal Organs (Hemoperitoneum) After Trauma, as Assessed by Focused Assessment With Sonography for Trauma (FAST), a Rapid Bedside Ultrasound Examination.
Description: Number of subjects screening positive for blood around the abdominal organs (hemoperitoneum) after trauma, as assessed by focused assessment with sonography for trauma (FAST), a rapid bedside ultrasound examination.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | FAST Examination After Right Sided Roll (FASTeR)
Number analyzed (Participants) | 182
Participants | 65

ADVERSE EVENTS:
Time Frame: At study visit, up to 24 hours
Arm/Group | FAST Examination After Right Sided Roll (FASTeR)
All-Cause Mortality (participants affected / at risk) | 0/182
Serious Adverse Events (participants affected / at risk) | 0/182
Other Adverse Events (participants affected / at risk) | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02991521/Prot_SAP_000.pdf